CLINICAL TRIAL: NCT01049841
Title: Phase I Study of Perifosine With Temsirolimus for Recurrent Pediatric Solid Tumors
Brief Title: Perifosine With Temsirolimus for Recurrent Pediatric Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: University of Wisconsin, Madison (Other); Duke University (Other); NATL COMP CA NETWORK (Unknown); Pfizer (Industry); AEterna Zentaris (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-124
Record Dates: First submitted 2010-01-14; First posted 2010-01-15 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-03

CONDITIONS: Pediatric Solid Tumors
Keywords: pediatric; children; perifosine; temsirolimus; recurrent; progressive; 09-124
MeSH Terms: conditions — Recurrence | interventions — perifosine; temsirolimus

ARMS (1):
- perifosine + temsirolimus (Experimental): This is a single arm, phase I study. Eligible patients will receive a loading dose of oral perifosine on the first day, followed by a maintenance dose starting on the second day until progression. Each patient is assigned to a group according to their body surface area (BSA). Temsirolimus will be combined with perifosine at four dose levels to determine the MTD for the combination therapy. Temsirolimus dosing will start on the same day as the perifosine load.
  Interventions: Drug: perifosine + temsirolimus

INTERVENTIONS:
Drug: perifosine + temsirolimus — The patient will take oral tablets of perifosine at a dose and frequency to be determined their height, weight and time when they enter the study as those entering early will be treated with lower dose levels (dosing frequency will vary from once a week to daily). The patient will receive an intravenous injection of temsirolimus once a week at a dose to be determined by their height, weight and time when they enter the study as those entering early will be treated with lower doses. In addition they will be asked to keep a medicine diary.

SUMMARY:
The purpose of this study is to test the safety and effectiveness of 2 drugs, perifosine in combination with temsirolimus in children with solid tumors. Neither drug is currently part of the standard treatment of solid tumors in children. Both drugs have been tested alone to treat solid tumors in children with little success. There is now new insight that if given together, perifosine and temsirolimus may work together to stop the growth of solid tumors and may also make them shrink. The doctor wants to find out what effects; good and/or bad, perifosine in combination with temsirolimus has on the patient and the cancer. The doctors are testing four different dose schedules of perifosine with temsirolimus and the patient will be asked to partake in one of the dose schedules. The dose schedule will be lower for those enrolled early in the study.

ELIGIBILITY:
Inclusion Criteria:

* Any solid tumor that has failed standard therapy
* Patient must have evidence of tumor by CT, MRI, MIBG scan, serum markers, or tissue sampling.
* Age ≤ 21 years (age ≤ 35 years for biopsy proven medulloblastoma or neuroblastoma)
* Karnofsky/Lansky performance status ≥ 50% (Karnofsky score for age> 16 years and Lansky score for age ≤ 16 years)
* ANC≥ 1000 at least 24 hours off GCSF
* Platelets ≥ 100K at least one week off platelet transfusions
* Hg≥ 8g/dL at least one week off PRBC transfusion
* AST ≤ 2 x the upper limit of normal
* ALT ≤ 2 x the upper limit of normal
* Total bilirubin ≤ 2.0 mg/dl
* Patients must have cholesterol level < 350 mg/dl and triglycerides level < 400 mg/dl because temsirolimus can induce hyperlipidemia.
* Serum creatinine ≤ 1.5 x the upper limit of normal for age, or calculated creatinine clearance or nuclear GFR ≥ 70 ml/min/1.73 m2.
* ≥ 3 weeks since last non-nitrosourea chemotherapy
* ≥ 6 weeks since last nitrosoureas
* ≥ 4 weeks since last RT
* Patients must agree to practice adequate contraception. Females of childbearing potential must have a negative serum B-HCG pregnancy test documented within 14 days prior to registration. Females must not be breast feeding.
* Patients must be able to swallow tablets whole
* Patients that participated in the phase I single agent perifosine study for recurrent pediatric solid tumors and did not experience a DLT are eligible to participate in this study and can start ≥ 2 weeks since last dose of perifosine
* Patients that have been previously treated with an mTOR inhibitor can still enroll in this trial as long as they did not experience a DLT in the single agent mTOR inhibitor trial

Exclusion Criteria:

* Pregnancy
* Patients must not have an uncontrolled active infection.
* HIV-Positive patients receiving combination anti-retroviral therapy are excluded from the study due to possible retro-viral drug interactions. HIV testing not required.
* Patients must not be taking EIAEDs. If patients were previously on EIAEDs that have been discontinued, patients must have been off the agent for at least 2 weeks prior to registration.
* History of or known pulmonary hypertension or history of or known pneumonitis.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of perifosine + temsirolimus combination in children with cancer. | 2 years

SECONDARY OUTCOMES:
To determine whether pharmacokinetic serum levels of both perifosine and temsirolimus correlate with toxicity. | 2 years
To record preliminary data on the efficacy of the perifosine + temsirolimus combination. | 2 years
If previously resected tissue is available, determine whether molecular features predict response including, Elevated PI3K/AKT/mTOR signaling, Elevated RAS/MAPK signaling, Cell cycle markers | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ira Dunkel, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Sun W, Modak S. Emerging treatment options for the treatment of neuroblastoma: potential role of perifosine. Onco Targets Ther. 2012;5:21-9. doi: 10.2147/OTT.S14578. Epub 2012 Mar 2. PMID 22419878
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org